CLINICAL TRIAL: NCT00496223
Title: A Phase I/II Study of Sunitinib and Dacarbazine in Patients With Metastatic Melanoma
Brief Title: A Phase I/II Study of Sunitinib and Dacarbazine
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: toxicities required dose reduction compromising effectiveness and PI left Moffitt
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Adil Daud, M.D., UCSF (formerly at H. Lee Moffitt Cancer Center & Research Institute)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14743
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Melanoma
Keywords: Sunitinib; Dacarbazine; Melanoma
MeSH Terms: conditions — Melanoma | interventions — Sunitinib; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Sunitinib; Drug: Dacarbazine

INTERVENTIONS:
Drug: Sunitinib — Sunitinib will be given PO once daily on days 1-14 of each 21 day cycle. The exact dose of sunitinib will be determined during the Phase I part of the trial.
Drug: Dacarbazine — Dacarbazine will be given at 1000 mg/m2 on day 1 of every 21 day cycle.
  Other Names: DTIC

SUMMARY:
This is a combination Phase I/II design that explores the toxicity and activity of Sunitinib and Dacarbazine (DTIC) for metastatic melanoma. The initial Phase I part of this trial will consist of a dose escalation of sunitinib while keeping the DTIC dose constant. If no DLT is seen, this dose will be the suggested Phase II trial dose. If less than 2 disease responses are seen, patients will not be enrolled any further, and the study will be considered negative for activity. If a clinical response is seen, patients will continue to be enrolled.

DETAILED DESCRIPTION:
This is a combination Phase I/II design that explores the toxicity and activity of a combination of sunitinib and Dacarbazine (DTIC) for metastatic melanoma. Screening tests (pre-study) will consist of a history, physical, CBC, CMP, EKG, pregnancy test for women of childbearing age, amylase (blood test for diagnoses of pancreatitis or other pancreatic diseases), staging CT, and PK. Also, on day 1, these tests will be repeated - a history, physical, toxicity assessment, CBC, and amylase test. Re-staging tests will be performed after 2 complete cycles and follow up as indicated clinically.

The initial Phase I part of this trial will consist of a dose escalation of sunitinib while keeping the DTIC dose constant. Sunitinib will be given 2 weeks on and 1 week off with DTIC given once every 21 days for one cycle. If no DLT is seen, the maximum tolerated sunitinib dose will be the suggested as the Phase II trial dose.

Tumor response will be measured after 2 complete cycles. Subsequently, during Phase II the trial will enroll more patients; if less than 2 responses are seen, patients will not be enrolled any further, and the study will be considered negative for activity. But, if a clinical response is seen, more patients will be enrolled at the Phase II dose.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented Stage IV or unresectable Stage III melanoma
* Resolution of all acute toxic effects of prior radiotherapy or surgical procedures to NCI CTCAE Version 3.0 grade less than or equal to 1
* Adequate organ function as defined by the following criteria:

  1. Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) less than or equal to 2.5 x local laboratory upper limit of normal (ULN), or AST and ALT less than or equal to 5 x ULN if liver function abnormalities are due to underlying malignancy
  2. Total serum bilirubin less than or equal to 1.5 x ULN
  3. Absolute neutrophil count (ANC) greater than or equal to 1500/mcL
  4. Platelets greater than or equal to 100,000/mcL
  5. Hemoglobin greater than or equal to 9.0 g/dL
  6. Serum calcium less than or equal to 12.0 mg/dL
  7. Serum creatinine less than or equal to 1.5 x ULN
* Patients with CNS metastasis must have had either:

  1. Resected CNS metastasis without evidence of recurrence for >12 weeks
  2. Brain metastasis treated by stereotactic radiosurgery without evidence of recurrence or progression for 12 weeks
  3. Multiple brain lesions treated with WBRT with stable disease off corticosteroids for at least 12 weeks prior to start of therapy
  4. Without any evidence of leptomeningeal disease
  5. Patients must be neurologically intact
* May have previous adjuvant therapy with interferon, vaccines or therapy with IL-2 or GM-CSF
* Measurable disease by RECIST criteria
* In the phase I part of the trial patients with evaluable but not measurable disease may be allowed with the permission of the PI
* ECOG PS 0-2

Exclusion Criteria:

* Major surgery or radiation therapy within 4 weeks of starting the study treatment.
* NCI CTCAE grade 3 hemorrhage within 4 weeks of starting the study treatment.
* History of or known carcinomatous meningitis, or evidence of symptomatic leptomeningeal disease on screening CT or MRI scan.
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
* Ongoing cardiac dysrhythmias of NCI CTCAE grade greater than or equal to 2.
* QTc >470 msec on baseline EKG.
* History of active CHF or LVEF<50% at screening echocardiogram.
* Hypertension that cannot be controlled by medications (>150/100 mm Hg despite optimal medical therapy).
* Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication.
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness or other active infection.
* Concurrent treatment on another clinical trial. Supportive care trials or non-treatment trials, e.g. QOL, are allowed.
* Ongoing treatment with therapeutic doses of Coumadin (low dose Coumadin up to 2 mg po daily for thromboembolism prophylaxis is allowed).
* Pregnancy or breastfeeding. Female subjects must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy. All female subjects with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment. Male subjects must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.
* Patients may not have had previous treatment with a DTIC or temozolomide based chemotherapy regimen. In the Phase II part of the trial patients may not have had treatment with any chemotherapy regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-09; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To determine the toxicity and safety of this combination and determine the recommended Phase II dose of this combination. | 6 months
To determine the overall response rate of the combination of sunitinib and DTIC as the first line treatment in stage IV malignant melanoma. | 4 months
To determine the progression free survival (PFS) of disease of patients treated with the combination of sunitinib and DTIC. | 2 years

SECONDARY OUTCOMES:
To determine Overall Survival of patients treated with this combination. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Adil Daud, M.D., Principal Investigator — UCSF (formerly at H. Lee Moffitt Cancer Center & Research Institute)
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials Website — http://www.moffitt.org